CLINICAL TRIAL: NCT05736653
Title: Strengthening Task Specific Activation of Paretic Hand Muscles After moderate-to- Severe Chronic Stroke
Brief Title: PCMS Task After Moderate-to-severe Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Amit Sethi, Associate Professor, University of Utah
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 00179089; R21HD108462 (NIH)
Record Dates: First submitted 2023-02-10; First posted 2023-02-21 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Stroke
Keywords: Stroke; Hand; Brain stimulation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: We will employ a single group pre-post design.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (6):
- Task-specific PCMS, PCMS-rest, Task-specific sham-PCMS (Experimental): During Task-specific paired corticospinal-motor neuronal stimulation (PCMS) participants will receive PCMS [Transcranial Magnetic Stimulation (TMS) + Peripheral Nerve Stimulation (PNS)] with task-specific practice.
  During PCMS rest participants will receive PCMS (TMS + PNS) without task-specific practice.
  During Task-specific sham-PCMS participants will receive task-specific practice with sham PCMS (TMS + PNS).
  Interventions: Device: Task-specific PCMS; Device: Task-specific sham-PCMS; Device: PCMS-rest
- Task-specific PCMS, Task-specific sham-PCMS, PCMS-rest (Experimental): During Task-specific PCMS participants will receive PCMS (TMS + PNS) with task-specific practice.
  During PCMS rest participants will receive PCMS (TMS + PNS) without task-specific practice.
  During Task-specific sham-PCMS participants will receive task-specific practice with sham PCMS (TMS + PNS).
  Interventions: Device: Task-specific PCMS; Device: Task-specific sham-PCMS; Device: PCMS-rest
- PCMS-rest, Task-specific PCMS, Task-specific sham-PCMS (Experimental): During Task-specific PCMS participants will receive PCMS (TMS + PNS) with task-specific practice.
  During PCMS rest participants will receive PCMS (TMS + PNS) without task-specific practice.
  During Task-specific sham-PCMS participants will receive task-specific practice with sham PCMS (TMS + PNS).
  Interventions: Device: Task-specific PCMS; Device: Task-specific sham-PCMS; Device: PCMS-rest
- PCMS-rest, Task-specific sham-PCMS, Task-specific PCMS (Experimental): During Task-specific PCMS participants will receive PCMS (TMS + PNS) with task-specific practice.
  During PCMS rest participants will receive PCMS (TMS + PNS) without task-specific practice.
  During Task-specific sham-PCMS participants will receive task-specific practice with sham PCMS (TMS + PNS).
  Interventions: Device: Task-specific PCMS; Device: Task-specific sham-PCMS; Device: PCMS-rest
- Task-specific sham-PCMS, Task-specific PCMS, PCMS-rest (Experimental): During Task-specific PCMS participants will receive PCMS (TMS + PNS) with task-specific practice.
  During PCMS rest participants will receive PCMS (TMS + PNS) without task-specific practice.
  During Task-specific sham-PCMS participants will receive task-specific practice with sham PCMS (TMS + PNS).
  Interventions: Device: Task-specific PCMS; Device: Task-specific sham-PCMS; Device: PCMS-rest
- Task-specific sham-PCMS, PCMS-rest, Task-specific PCMS (Experimental): During Task-specific PCMS participants will receive PCMS (TMS + PNS) with task-specific practice.
  During PCMS rest participants will receive PCMS (TMS + PNS) without task-specific practice.
  During Task-specific sham-PCMS participants will receive task-specific practice with sham PCMS (TMS + PNS).
  Interventions: Device: Task-specific PCMS; Device: Task-specific sham-PCMS; Device: PCMS-rest

INTERVENTIONS:
Device: Task-specific PCMS — 120 pairs of TMS and PNS volleys will be administered during electromyography-triggered functional electrical stimulation (FES)-assisted task-specific training (task-specific PCMS). In the task-specific PCMS, participants will first grasp a spherical ball when prompted by an auditory 'Ready' cue, and upon seeing a visual 'Go' cue will voluntarily extend the wrist and fingers to release the ball. After the 'Go cue', our customized stimulation delivery algorithm triggers the TMS and PNS only when the extensor digitorum communis (EDC) muscle activity exceeds a pre-determined threshold. The algorithm will then trigger FES to EDC after detecting EDC activity (~2 ms after PNS) for the next 2 seconds, allowing the pairing of PCMS (TMS and PNS) with the voluntary movement of EDC without the confounding effects of FES.
Device: Task-specific sham-PCMS — 120 pairs of sham-PCMS stimuli will be administered during task-specific practice. The TMS coil will be placed ~10 cm behind the participant's head, and PNS electrodes will be placed in the same position as for task-specific PCMS, but no stimulation will be delivered. Like the task-specific PCMS condition, participants will perform the same grasp and release a ball task in an identical manner. FES will be delivered after detecting voluntary EDC activity, similar to the task-specific PCMS condition.
Device: PCMS-rest — 120 pairs of TMS and PNS volleys will be administered with the EDC muscle at rest every 10 s (~20 min, 0.1 Hz). TMS will be used to elicit motor-evoked potentials (MEPs). Antidromic activation of spinal motor neurons will be elicited by supramaximal peripheral nerve stimulation (PNS) applied to the radial nerve near the elbow. Volleys will be timed to arrive in the spinal cord based on central and peripheral conduction times calculated for each subject so that the pre-synaptic terminal is depolarized via TMS ~1-2 ms before spinal motor neurons are depolarized via PNS at a pulse duration of 200us. We will also perform stimulation of the cervical roots (C-root) by placing the coil behind the neck and stimulating the C-root (C6 and C7 vertebrae), which innervate the finger extensor muscles. Conduction times will be calculated from latencies of the primary motor area (M1) MEP, C-root, and M-wave.

SUMMARY:
Researchers at the University of Pittsburgh are conducting a research study to see how combining brain, nerve, and hand stimulation affect hand movement after stroke. The primary purpose of this study is to examine changes in the connection between the brain and the weak hand muscles after the combined brain, nerve, and hand stimulation. The primary hypothesis is that the combined brain, nerve, and hand stimulation will increase the the connection between the brain and the weak hand muscles. The secondary purpose of this study is to examine changes in weak hand's movement and function after the combined brain, nerve, and hand stimulation. The secondary hypothesis is that the combined brain, nerve, and hand stimulation will increase weak hand movement and function.

DETAILED DESCRIPTION:
A total of 40 participants will be enrolled in this study. During the intervention sessions, Participants will receive three combinations of the brain, hand, and nerve stimulations.

Each participant will complete three intervention sessions for the short-term effect of the intervention. The time between sessions is 3-7 days. After data collection is completed for the short-term effect part of the study, 5 out of 40 participants will be randomly chosen to enroll in the long-term effect part of the intervention. Those participants will take part in 18 intervention sessions. The sessions will be administered three times a week for six weeks.

In the short-term effect part of the study, participants will complete the following three sessions:

1. Repeated brain, hand, and nerve stimulations while practicing a task. In this session, participants will receive 120 pairs of brain, hand, and nerve stimulation while repeatedly grasp and release a ball with the weak hand. The hand stimulation will help participants to release the ball.
2. Repeated brain and nerve stimulations during rest. In this session, participants will receive 120 pairs of brain and nerve stimulation while the weak hand is resting (or not performing a task).
3. Hand stimulation while practicing a task. In this session, participants will practice grasping and releasing the task 120 times with hand stimulation. The hand stimulation will help participants to release the ball.

In the long-term effect part of the study, participants will complete the following session (3/week for 6 weeks):

During the intervention, participants will receive repeated brain, hand, and nerve stimulations while practicing a task. They will receive 120 pairs of brain, hand, and nerve stimulation while repeatedly grasp and release a ball with the weak hand. The hand stimulation will help participants to release the ball. We will give rest breaks during the practice of the task.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-85 years
2. Diagnosis of first-ever subcortical stroke (single cerebrovascular accident)
3. Stroke onset of at least six months prior to the time of participation
4. A score of at least 1 out of 2 on the spherical grasping item of the Fugl-Meyer Upper Extremity Subscale to allow participants to grasp the ball
5. Cognitive skills to actively participate, as indicated by scores of > 23 on the Mini-Mental Status Examination
6. English speaking

Exclusion Criteria:

1. Inability to elicit a motor evoked potential (MEP) in the EDC muscle even with a 20% background muscle contraction
2. Presence of severe aphasia
3. Excessive spasticity of the wrist and finger muscles, defined as a Modified Ashworth Score >2
4. Diagnosis of neurological disorders other than stroke
5. History of seizure or epilepsy
6. Orthopedic/musculoskeletal conditions (e.g., arthritis) affecting the upper extremity
7. Presence of metallic implants in the head or neck
8. Currently or planning to become pregnant
9. Difficulty maintaining alertness or remaining still
10. Ferromagnetic metallic implants, pacemakers, other implanted devices, or ventilators for magnetic resonance imaging (MRI)
11. Bodyweight > 300 lbs due to MRI scanner dimensions (for subjects also undergoing MRI)
12. Psychiatric diagnosis according to the criteria of the Diagnostic and Statistical Manual of Mental Disorder, Fifth Edition (DSM-V), or who are on psychotropic medication
13. Life expectancy less than the duration of the study
14. Excessive pain in the paretic hand, defined as a Visual Analog Scale Score >4
15. Participation in concurrent occupational therapy
16. Current use of recreational drugs and stimulants like cocaine and methylenedioxymethamphetamine (MDMA)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-29 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Transcranial magnetic stimulation to evaluate corticospinal transmission | Change from baseline up to 30-minutes post intervention
  Corticospinal transmission will be assessed by examining the percent change of the peak-to-peak motor evoked potential (MEP) amplitude relative to baseline.

SECONDARY OUTCOMES:
Voluntary force production to evaluate motor performance | Change from baseline up to 30-minutes post intervention
  We will measure force production of the wrist and finger extensors (EDC) to evaluate motor performance using load cells embedded in cushioned customized platforms. Participants will perform isometric wrist and finger extension movements against load cells. We will calculate the percent change of maximum force output.
Maximum finger excursions to evaluate motor performance | Change from baseline up to 30-minutes post intervention
  Three-dimensional biomechanical data will be collected to evaluate motor performance using a motion capture system. Reflective markers will be placed on the participant's paretic forearm, hand, and fingers to track wrist and finger movements during a maximum hand opening task. Hand biomechanics will be evaluated by computing the percent change of maximum finger excursions during the hand opening task.
Maximum finger spread to evaluate motor performance | Change from baseline up to 30-minutes post intervention
  Three-dimensional biomechanical data will be collected to evaluate motor performance using a motion capture system. Reflective markers will be placed on the participant's paretic forearm, hand, and fingers to track wrist and finger movements during a maximum hand opening task. Hand biomechanics will be evaluated by computing the percent change of maximum finger spread during the hand opening task.
Box and Block Test | Change from baseline up to 30-minutes post intervention
  The Box and Block Test (BBT) measures unilateral gross manual dexterity and the ability to release objects. We will calculate the percent change of the total number of blocks transferred in one minute.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Sethi, PhD, Principal Investigator — University of Utah
Locations (1):
- Neural Plasticity Rehabilitation and Movement Dynamics Lab, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No